CLINICAL TRIAL: NCT03373734
Title: Feasibility Study Investigating the Efficacy and Acceptability of a Pregnancy Focussed Online Cognitive Behavioural Therapy Package: Enjoy Your Bump
Brief Title: Enjoy Your Bump : Online Cognitive Behavioural Therapy in Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: Edinburgh & Lothians Health Foundation (Unknown); Tommy's Edinburgh Maternal & Fetal Health Centre (Unknown); National Health Service (NHS) Lothian (Unknown); Five Areas Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: AC17015
Record Dates: First submitted 2017-10-11; First posted 2017-12-14 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Perinatal Mental Health; Antenatal Depression; Antenatal Anxiety
Keywords: Online Cognitive Behavioural Therapy; Pregnancy; Self-help

STUDY DESIGN:
Intervention Model Description: Enjoy Your Bump is an online life skills course based on cognitive behavioural therapy principles. It has been designed to address issues pertinent to mood in pregnancy. The course compiles five modules delivered in the form of an online slideshow with audio. It can be accessed from a range of devices. There are a series of worksheets the user can access and download which accompany the modules.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Enjoy Your Bump — Online life skills course based on Cognitive Behavioural Therapy Principles.
  Other Names: Five Areas Ltd Enjoy Your Bump

SUMMARY:
A feasibility study evaluating how acceptable women experiencing low mood or anxiety during their pregnancy find an online Cognitive Behavioural Therapy course called 'Enjoy Your Bump'. This project will also begin to explore the effectiveness of this programme as a low intensity self-help intervention for mild to moderate depressive symptoms during pregnancy.

DETAILED DESCRIPTION:
'Enjoy Your Bump (EYB)' is an online life skills course based on Cognitive Behavioural Therapy (CBT) principles which has been designed to specifically support women in the antenatal period. A survey of women and health professionals has demonstrated that this is a resource that both groups find acceptable. The aim of this quasi-experimental feasibility study is to evaluate the user experience and efficacy of this online programme as a non-pharmacological, low intensity intervention for women experiencing mild-moderate depressive symptoms in pregnancy. This will be achieved by measuring depression and anxiety as well as measures of attachment to the developing baby, pre and post intervention. It is hoped the results from this study will help inform whether this is a resource that should be made more widely available to women in the National Health Service (NHS). It is hypothesised that the 'Enjoy Your Bump' will be an acceptable and effective intervention for women experiencing mild to moderate depressive symptoms in the antenatal period.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Mild-moderate chronic perinatal mental health identified by a score of 2 or higher on PHQ-2 and/or GAD-2.
* 16+0 to 32+6 weeks at recruitment

Exclusion Criteria:

* Severe perinatal mental health problem such as schizophrenia, bipolar disorder, substance abuse/dependence, active risk of self-harm.
* Already receiving psychological therapy.
* Insufficient English language to engage with intervention or complete questionnaires.
* Unable to give informed consent.
* Illiterate
* No internet access
* Taking part in another current research project focused on mental health.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of recruitment and retention. | Measured at 12 months post study start date
  Evaluate how many women are recruited to the study, how many women complete the online modules and how many women give feedback on their experience via an online questionnaire.
Evaluation of feedback questionnaire data. | Measured at 12 months post study start date
  Evaluate the qualitative feedback women give regarding their experience of the intervention using an online questionnaire.
Estimation of effect size for changes in depression. | Measured at 12 months post study start date.
  Obtain an estimate of effect size for changes in depression, from pre to post intervention.
  Change in effect size for depression will be measured using Standardised Mean Difference (SMD) of scores on Patient Health Questionnaire-9 (PHQ-9) from pre to post intervention.
Estimate of Effect Size for changes in depression (2) | Measured at 12 months post study start date.
  Obtain an estimate of effect size for changes in depression, from pre to post intervention.
  Change in effect size for depression will be measured using Standardised Mean Difference (SMD) of scores on the Warwick Edinburgh Mental Wellbeing Scale (WEMWBS) from pre to post intervention.
Estimate of effect size for changes in depression (3) | Measured at 12 months post study start date.
  Obtain an estimate of effect size for changes in depression, from pre to post intervention.
  Change in effect size for depression will be measured using Standardised Mean Difference (SMD) of scores on the Edinburgh Postnatal Depression Score (EPDS) from pre to post intervention.
Estimation of effect size for changes in anxiety. | Measured at 12 months post study start date.
  Effect size for Anxiety will be measured using SMD for Generalised Anxiety-7 questionnaire scores before and after intervention.
Estimation of effect size for changes in social function. | Measured at 12 months post study start date.
  Effect size for social function will be measured using SMD for score on pregnancy experience scale (PES) pre and post intervention.
Estimation of effect size for changes in attachment. | Measured at 12 months post study start date.
  Effect size in attachment will be measured using SMD for scores on Prenatal Attachment Inventory both before and after intervention.

SECONDARY OUTCOMES:
Depression score (1) | Scores will be recorded at recruitment to study (between 16 - 32+6 weeks gestation), Post Enjoy Your Bump Intervention (before 38 weeks gestation) and 12 weeks Postnatal.
  Measure depression pre and post intervention using a standardised assessment tool:
  Patient Health Questionnaire-9 (PHQ-9). This standardised questionnaire measures depression. Score ranges 0-27 with 0 representing least depressed and 27 representing most depressed.
Depression score (2) | Scores will be recorded at recruitment to study (between 16 - 32+6 weeks gestation), Post Enjoy Your Bump Intervention (before 38 weeks gestation) and 12 weeks Postnatal.
  Measure depression pre and post intervention using standardised assessment tool:
  Edinburgh Postnatal Depression Score (EPDS). Another standardised questionnaire. Scores range from 0-30. '0' represents least depressed and '30' represents most depressed.
Depression score (3) | Scores will be recorded at recruitment to study (between 16 - 32+6 weeks gestation), Post Enjoy Your Bump Intervention (before 38 weeks gestation) and 12 weeks Postnatal.
  Measure depression pre and post intervention using standardised assessment tool:
  . Warwick Edinburgh Mental Wellbeing Scale (WEMWS). Another standardised assessment of mood. Scores range from 14 - 70. '14' represents most depressed and '70' represents least depressed.
Anxiety score | Scores will be recorded at recruitment to study (between 16 - 32+6 weeks gestation), Post Enjoy Your Bump Intervention (before 38 weeks gestation) and 12 weeks Postnatal.
  Measure anxiety pre and post intervention using standardised assessment tool Generalised Anxiety Disorder-7 Item scale (GAD-7). This standardised questionnaire gives a score between '0-21'. '0' represents the least anxious and '21' represents the most anxious.
Pregnancy Experience | Scores will be recorded at recruitment to study (between 16 - 32+6 weeks gestation), Post Enjoy Your Bump Intervention (before 38 weeks gestation)
  Measure pregnancy experience pre and post intervention using the Pregnancy Experience Scale (PES). This 41-item questionnaire measures participants feelings towards social issues related to their pregnancy. Total score ranges from 0-123. '0' represents no negative feelings towards experience in pregnancy and '123' represents maximum negative experience towards experience of pregnancy.
Measure mother-baby relationship (Antenatal) | Scores will be recorded at recruitment to study (between 16 - 32+6 weeks gestation), and Post Enjoy Your Bump Intervention (before 38 weeks gestation)
  Evaluate the mother-baby attachment in the antenatal period pre and post intervention using the Prenatal Attachment Inventory (PAI)
  The Prenatal Attachment Inventory is a 21-item questionnaire with scores ranging from 21-84 with '21' representing most attached and '84' the least attached.
Measure mother-baby relationship (Postnatal) | Score recorded at 12 weeks postnatal
  Evaluate the mother-baby attachment post intervention in the postnatal period using The Maternal Attachment Inventory (MAI).
  The Maternal Attachment Inventory is a 26-item questionnaire. Total ranges from '26-104'. 26 represents poor attachment and 104 represents good attachment.
Time taken to complete intervention (1) | Data will be recorded at participant completion of Enjoy Your Bump intervention. Participants are required to complete intervention before they are 38+0 weeks pregnant.
  Quantify how long it typically takes participants to complete the intervention.
  This will be assessed in 'minutes participant spent active using the intervention'. This data in recorded on the online programme for researcher to see. We will also measure in weeks, how long it took participants to complete all 5 modules of the Enjoy Your Bump intervention.
Time taken to complete intervention (2). | Data will be recorded at participant completion of Enjoy Your Bump intervention. Participants are required to complete intervention before they are 38+0 weeks pregnant.
  Quantify how long it typically takes participants to complete the intervention. We will measure in weeks and days, how long it took participants to complete all 5 modules of the Enjoy Your Bump intervention from recruitment date.
Delivery and support of intervention | Data will be recorded at participant completion of Enjoy Your Bump intervention. Participants are required to complete intervention before they are 38+0 weeks pregnant.
  Test and evaluate the ability to deliver and support the intervention. This will be measured by asking participants in the evaluation questionnaire to comment on how they evaluated the support they received.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca M Reynolds, PHD, Principal Investigator — University of Edinburgh
Locations (1):
- NHS Lothian / University of Edinburgh, Edinburgh, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2017-07-05): https://cdn.clinicaltrials.gov/large-docs/34/NCT03373734/Prot_000.pdf
  • Informed Consent Form (2017-07-05): https://cdn.clinicaltrials.gov/large-docs/34/NCT03373734/ICF_001.pdf